CLINICAL TRIAL: NCT05133882
Title: A Phase Ib/II, Multi-center, Open Clinical Trial of Crifortinib Besylate Combined With Chemotherapy in Newly-treated Adult Subjects With Acute Myeloid Leukemia
Brief Title: A Phase Ⅰb/Ⅱ Clinical Study of Clifutinib Besylate Combined With Chemotherapy in the Treatment of Newly Diagnosed AML
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: PCD-DHEC73543-16-002
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Arm 1:30 mg Arm 2:40 mg Arm 3:60 mg
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Experimental): Queue 1:Clifutinib Besylate:30mg qd d8-21;Daunorubicin 60 mg/m2 qd d1-3;Cytarabine 100 mg/m2 qd d1-7 Queue 1:Clifutinib Besylate:30mg qd d1-28 ;Azacitidine 75 mg/m2 qd d1-7
  Interventions: Drug: Clifutinib Besylate
- Arm 2 (Experimental): Queue 1:Clifutinib Besylate:40mg qd d8-21;Daunorubicin 60 mg/m2 qd d1-3;Cytarabine 100 mg/m2 qd d1-7 Queue 1:Clifutinib Besylate:40mg qd d1-28 ;Azacitidine 75 mg/m2 qd d1-7
  Interventions: Drug: Clifutinib Besylate
- Arm 3 (Experimental): Queue 1:Clifutinib Besylate:60mg qd d8-21;Daunorubicin 60 mg/m2 qd d1-3;Cytarabine 100 mg/m2 qd d1-7 Queue 1:Clifutinib Besylate:60mg qd d1-28 ;Azacitidine 75 mg/m2 qd d1-7
  Interventions: Drug: Clifutinib Besylate

INTERVENTIONS:
Drug: Clifutinib Besylate — The queue 1 is divided into Induction therapy and Consolidation therapy and Maintenance treatment The queue 2 will receive oral Clifutinib Besylate once daily until disease progression or unacceptable toxicity occurs
  Other Names: HEC73543

SUMMARY:
This is a multi-center open clinical study aimed at evaluating the efficacy and safety of Clifutinib Besylate combined with chemotherapy in newly-treated adult subjects with AML

DETAILED DESCRIPTION:
Main purpose:To evaluate the tolerability and safety of Clifutinib Besylate combined with DA (Cytarabine + Daunorubicin) or AZA (Azacitidine) in newly-treated adult AML subjects; explore reasonable therapeutic doses through climbing tests in different dose groups.

To evaluate the efficacy of Clifutinib Besylate combined with DA or AZA in newly treated adult AML subjects.

Secondary purpose:To observe the pharmacokinetic (PK) characteristics of Clifutinib combined with DA or AZA in newly-treated adult AML subjects and the drug interaction between Clifutinib and AZA at the same time.Observe the correlation of different subtypes and prognostic risk with the efficacy of Clifutinib and the changes of genes before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1.Cohort 1: 18 years old ≤ age ≤65 years old;Cohort 2: The dose escalation trial only included AML subjects aged ≥60 years; the extended trial included subjects who were ≥60 years old or between 18 and 59 years old (including 18 and 59 years old) and could not tolerate strong chemotherapy.

  2.It can be primary AML or AML secondary to MDS, and has not been treated; the extension phase requires the subject to be positive for the FLT3-ITD mutation.

  3.The ECOG score according to the requirements of different groups is as follows: Cohort 1: 0~1 points; Cohort 2: Age ≥60 years old: 0~2 points; Age 18~59 years old (including 18 and 59 years old): 0~3 points.

  4.Expected survival time ≥ 12 weeks. 5. Subjects must have adequate organ function. 6.subjects voluntarily participated in the study, and signed a written informed consent form by themselves or their guardians.

Exclusion Criteria:

* 1.Diagnosed as APL and manifested as t(15;17)(q22;q12) chromosomal translocation, or BCR-ABL positive leukemia；Diagnosed as secondary to AML due to previous chemotherapy or radiotherapy of other tumors; previously received FLT3 inhibitor.

  2.AML secondary to myeloproliferative tumor (MPN) or acute lymphoblastic leukemia (ALL).

  3.Subjects who have infiltrated the central nervous system in the past or present.

  4.Concomitant with other malignant tumors within 5 years before the first medication.

  5.Thrombosis or embolism occurred within 12 months before the first medication. 6.Pulmonary function tests indicate that subjects have DLCO ≤50% or FEV1 ≤60%, or have difficulty breathing during rest or require continuous oxygen inhalation.

  7.Subjects with uncontrollable, active infections。 8.Clinically obvious gastrointestinal abnormalities, which may affect the intake, transport or absorption of drugs (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.), or subjects undergoing total gastrectomy。 9.Subjects with a history of psychotropic drug abuse and unable to quit or those with mental disorders。 10.Researchers believe that those who have other severe acute or chronic diseases who are not suitable for participating in clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose(MTD) | day 1-28
  Safety and Tolerability assessed through adverse events to determine maximum tolerated dose
Composite CR rate | Up to 12 months
  CR + CRi +CRMRD-

SECONDARY OUTCOMES:
Duration of response | up to 12 months
  The time from receive CR / CRi/CRMRD-/PR to relapse
Objective response rate | up to 12 months
  CR + CRi +CRMRD- + PR
Event Free Survival | up to 12 months
  From the first time taking experimental drug to treatment failure or progression or relapse or death
Overall Survival | up to 12 months
  From the first time taking experimental drug to death

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, Doctor, Study Chair — First Affiliated Hospital of Zhejiang University
Locations (1):
- the First Affiliated Hospital,College of Medicine,Zhejiang University, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No